CLINICAL TRIAL: NCT02749994
Title: A Clinical Trial to Compare the Efficacy and Safety of a Combination Therapy of Ezetimibe and Rosuvastatin Versus Monotherapy of Rosuvastatin in Hypercholesterolemia Patients (I-ROSETTE Study)
Acronym: I-ROSETTE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: ID-ROEZ-302
Record Dates: First submitted 2016-04-19; First posted 2016-04-25 (Estimated); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Rosuvastatin Calcium; Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- R5 (Active Comparator): Rosuvastatin 5mg
  Interventions: Drug: Rosuvastatin
- R10 (Active Comparator): Rosuvastatin 10mg
  Interventions: Drug: Rosuvastatin
- R20 (Active Comparator): Rosuvastatin 20mg
  Interventions: Drug: Rosuvastatin
- R5/E10 (Experimental): Rosuvastatin 5mg/Ezetimibe 10mg
  Interventions: Drug: Rosuvastatin; Drug: Ezetimibe
- R10/E10 (Experimental): Rosuvastatin 10mg/Ezetimibe 10mg
  Interventions: Drug: Rosuvastatin; Drug: Ezetimibe
- R20/E10 (Experimental): Rosuvastatin 20mg/Ezetimibe 10mg
  Interventions: Drug: Rosuvastatin; Drug: Ezetimibe

INTERVENTIONS:
Drug: Rosuvastatin
Drug: Ezetimibe
  Arms: R10/E10; R20/E10; R5/E10

SUMMARY:
A phase Ⅲ, multi-center, randomized, double-blinded, active comparator, factorial design clinical trial to compare the efficacy and safety of a combination therapy of ezetimibe and rosuvastatin versus monotherapy of rosuvastatin in hypercholesterolemia patients.

ELIGIBILITY:
Inclusion Criteria:

1. 19 ~ 79 years old
2. Patients who confirmed hypercholesterolemia.
3. Patients who requiring drug therapy according to NCEP ATP(National Cholesterol Education Program Adult Treatment Panel) III Guideline at Visit2.
4. Patients with Triglyceride< 400 at Visit 2.
5. Patients who have a wash-out period over 4 weeks for other drugs that can affect lipid profile.(Patients who have lipid regulators should have washout period over six weeks)
6. Patients who agreed to participate in the trial

Exclusion Criteria:

1. Patients who have a history of myopathy or rhabdomyolysis by statin treatment or hypersensitivity to statin HMG CoA(3-hydroxy-3-methylglutaryl-coenzyme) reductase inhibitors) or ezetimibe.
2. A heavy alcohol consumer. (alcohol > 25 units/week)
3. Patients with severe renal disease. (creatinine ≥ 2.0 mg/dL)
4. Patients with active liver disease and AST(aspartate transaminase) or ALT(alanine transaminase) > 2 times of upper limit of normal range.
5. Patients with CPK(creatine phosphokinase) > 2 x upper limit of normal range.
6. Patients who have a endocrine or metabolic diseases known to affect the serum phospholipid or lipoprotein.
7. Patients with HIV(human immunodeficiency virus positive.
8. Patients who have a acute arteriopathy.
9. Patients with uncontrolled hypertension.
10. Patients who have hereditary problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption.
11. Patients who have a drugs absorption disorder by gastrointestinal surgery or gastrointestinal disorder.
12. Patients with tumor.
13. Patients who have hormonal therapy.
14. Pregnancy or breastfeeding patients who don't agree to use adequate contraception.
15. Patients who are judged unsuitable to participate in this study by investigator.
16. Patients taking other clinical trial drugs within 30 days from the time of visit for screening.

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2016-04; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline to 8 week in LDL-Cholesterol | baseline and 8 week

SECONDARY OUTCOMES:
Percent change from baseline to 4 and 8 week in Total Cholesterol | baseline to 4 and 8 week
Percent change from baseline to 4 and 8 week in Triglyceride | baseline to 4 and 8 week
Percent change from baseline to 4 and 8 week in HDL-Cholesterol | baseline to 4 and 8 week
Percent change from baseline to 4 and 8 week in non-HDL-Cholesterol | baseline to 4 and 8 week
Percent change from baseline to 4 and 8 week in Apolipoprotein B | baseline to 4 and 8 week
Percent change from baseline to 4 and 8 week in Apolipoprotein A1 | baseline to 4 and 8 week
Percent change from baseline to 4 week in LDL-Cholesterol | baseline to 4 week
Percent change from baseline to 4 and 8 week in hs-CRP(high-sensitivity C-reactive protein) | baseline to 4 and 8
The change of LDL-Cholesterol/HDL-Cholesterol ratio | baseline to 4 and 8 week
The change of Total Cholesterol/HDL-Cholesterol ratio | baseline to 4 and 8 week
The change of non-HDL-Cholesterol/HDL-Cholesterol ratio | baseline to 4 and 8 week
The change of Apolipoprotein B/Apolipoprotein A1 ratio | baseline to 4 and 8 week
The ratio of subjects who reach the goal of LDL-Cholesterol according to NCEP(National Cholesterol Education Program Adult Treatment Panel) III Guideline | baseline to 4 and 8 week

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-soo Kim, MD/PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hong SJ, Jeong HS, Ahn JC, Cha DH, Won KH, Kim W, Cho SK, Kim SY, Yoo BS, Sung KC, Rha SW, Shin JH, Han KR, Chung WS, Hyon MS, Lee HC, Bae JH, Rhee MY, Kwan J, Jeon DW, Yoo KD, Kim HS. A Phase III, Multicenter, Randomized, Double-blind, Active Comparator Clinical Trial to Compare the Efficacy and Safety of Combination Therapy With Ezetimibe and Rosuvastatin Versus Rosuvastatin Monotherapy in Patients With Hypercholesterolemia: I-ROSETTE (Ildong Rosuvastatin & Ezetimibe for Hypercholesterolemia) Randomized Controlled Trial. Clin Ther. 2018 Feb;40(2):226-241.e4. doi: 10.1016/j.clinthera.2017.12.018. PMID 29402522